CLINICAL TRIAL: NCT01129635
Title: Real-Time Intracardiac Impedograms of Left Ventricular Leads to Locate Sites of Latest Mechanical Delay in Cardiac Resynchronization Therapy
Brief Title: Optimal Coronary Sinus Lead Implantation Using Intracardiac Impedography and Magnetic Resonance Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Michael S. Lloyd, PI, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00036655; ACTSI-EP-001 (Other: Other)
Record Dates: First submitted 2010-05-05; First posted 2010-05-24 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Heart Failure, Systolic; Left Bundle Branch Block
Keywords: Heart failure; Cardiac resynchronization therapy; Regional left ventricular dyssynchrony; CRT
MeSH Terms: conditions — Heart Failure, Systolic; Bundle-Branch Block; Heart Failure | interventions — Cardiac Resynchronization Therapy; Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CRT Candidate (Experimental): Patients with NYHA Class III or IV heart failure; EF ≤ 30% and QRS duration ≥ 120 ms, who are scheduled for CRT surgery.
  Intervention: Cardiac Resynchronization Therapy (CRT) implantation
  Interventions: Procedure: Cardiac Resynchronization Therapy (CRT) implantation

INTERVENTIONS:
Procedure: Cardiac Resynchronization Therapy (CRT) implantation — The impedance measurement is performed during device implantation following CMR. After the RV and LV leads are inserted, secured and tested, they will be connected to the impedance monitor. Impedance recording of at least ten beats will be acquired and stored for future analysis. Each recording will be tagged with the anatomical location of the LV lead. Subsequently, the LV lead will be moved to a different location and the same procedure will be repeated until accessible coronary sinus sites are exhausted. The ultimate LV lead location is determined by the implanting electrophysiologist and is not constrained by the study protocol. Finally, the LV lead will be tested again and the rest of the implantation procedure will proceed as routine.
  Arm: CRT Candidate

SUMMARY:
Despite the dramatic effect of cardiac resynchronization therapy (CRT) on survival and morbidity in people with congestive heart failure, 50-70% of eligible patients do not respond to this intervention. There is retrospective evidence that placement of the left ventricular (LV) lead at the region of latest mechanical delay markedly improves response to CRT. However, there is no feasible way to gauge dyssynchrony at LV lead sites during CRT implantation. Impedance recordings from pacing lead tips allow for real-time assessment of mechanical motion and may represent a useful intraoperative tool to guide optimum placement of the LV lead during CRT implantation. This pilot trial will assess the use of intraoperative impedograms in humans to measure regional dyssynchrony at potential LV lead locations during CRT implantation.

DETAILED DESCRIPTION:
This is a clinical trial using intracardiac impedance signals (impedograms) to assess regional dyssynchrony at various sites of left ventricular (LV) lead placement in humans undergoing CRT device implantation. This study will test the following hypotheses during the funding period:

1. LV lead impedograms as an implant tool to place leads at sites of latest mechanical delay are feasible and correlate with other means of assessing dyssynchrony.
2. LV lead impedograms vary significantly depending on LV lead location.
3. There are several characteristics of LV lead impedograms that correlate with mechanical phenomena of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NYHA class III or IV heart failure
* LVEF ≤ 30%
* QRS duration ≥ 120 ms

Exclusion Criteria:

* Not a candidate for CRT implantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-06; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Anatomic correlation between largest Ts (see description) and site of longest delay among probed locations in the CMR dyssynchrony map. | Acute intraoperative measurement
  Parameter will be recorded for at least 10 consecutive heartbeats during sinus and RV paced rhythm
  Ts = The average time from the sensed RV IEGM to the peak of the LV impedance curve

SECONDARY OUTCOMES:
Differential correlation of Ts, Tp, and Td (see description) to the CMR dyssynchrony map. | Acute intraoperative measurement
  Ts: The average time from the sensed RV IEGM to the peak of the LV impedance curve.
  Tp: The average time from the paced RV IEGM to the peak of the LV impedance curve.
  Td: The difference between Ts and Tp (Tp - Ts).

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Lloyd, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Background] Abraham WT, Fisher WG, Smith AL, Delurgio DB, Leon AR, Loh E, Kocovic DZ, Packer M, Clavell AL, Hayes DL, Ellestad M, Trupp RJ, Underwood J, Pickering F, Truex C, McAtee P, Messenger J; MIRACLE Study Group. Multicenter InSync Randomized Clinical Evaluation. Cardiac resynchronization in chronic heart failure. N Engl J Med. 2002 Jun 13;346(24):1845-53. doi: 10.1056/NEJMoa013168. PMID 12063368
- [Background] Jessup M. MADIT-CRT--breathtaking or time to catch our breath? N Engl J Med. 2009 Oct 1;361(14):1394-6. doi: 10.1056/NEJMe0907335. Epub 2009 Sep 1. No abstract available. PMID 19723700
- [Background] Moss AJ, Hall WJ, Cannom DS, Klein H, Brown MW, Daubert JP, Estes NA 3rd, Foster E, Greenberg H, Higgins SL, Pfeffer MA, Solomon SD, Wilber D, Zareba W; MADIT-CRT Trial Investigators. Cardiac-resynchronization therapy for the prevention of heart-failure events. N Engl J Med. 2009 Oct 1;361(14):1329-38. doi: 10.1056/NEJMoa0906431. Epub 2009 Sep 1. PMID 19723701
- [Background] Couri DM, Mankad S. Cardiac resynchronization therapy. Curr Treat Options Cardiovasc Med. 2008 Dec;10(6):538-48. doi: 10.1007/s11936-008-0046-5. PMID 19026184
- [Background] Lloyd MS, Heeke S, Lerakis S, Langberg JJ. Reverse polarity pacing: the hemodynamic benefit of anodal currents at lead tips for cardiac resynchronization therapy. J Cardiovasc Electrophysiol. 2007 Nov;18(11):1167-71. doi: 10.1111/j.1540-8167.2007.00943.x. PMID 17764446
- [Background] Mounsey JP, Knisley SB. Anodal capture, cathodal capture, and left ventricular cardiac excitation. J Cardiovasc Electrophysiol. 2009 Jun;20(6):650-2. doi: 10.1111/j.1540-8167.2008.01418.x. Epub 2009 Jan 9. No abstract available. PMID 19175447
- [Background] Theis C, Bavikati VV, Langberg JJ, Lloyd MS. The relationship of bipolar left ventricular pacing stimulus intensity to cardiac depolarization and repolarization in humans with cardiac resynchronization devices. J Cardiovasc Electrophysiol. 2009 Jun;20(6):645-9. doi: 10.1111/j.1540-8167.2008.01378.x. Epub 2009 Dec 15. PMID 19207760
- [Background] Becker M, Franke A, Breithardt OA, Ocklenburg C, Kaminski T, Kramann R, Knackstedt C, Stellbrink C, Hanrath P, Schauerte P, Hoffmann R. Impact of left ventricular lead position on the efficacy of cardiac resynchronisation therapy: a two-dimensional strain echocardiography study. Heart. 2007 Oct;93(10):1197-203. doi: 10.1136/hrt.2006.095612. Epub 2007 Feb 19. PMID 17309913
- [Background] Becker M, Kramann R, Franke A, Breithardt OA, Heussen N, Knackstedt C, Stellbrink C, Schauerte P, Kelm M, Hoffmann R. Impact of left ventricular lead position in cardiac resynchronization therapy on left ventricular remodelling. A circumferential strain analysis based on 2D echocardiography. Eur Heart J. 2007 May;28(10):1211-20. doi: 10.1093/eurheartj/ehm034. Epub 2007 Apr 10. PMID 17426079
- [Background] Chung ES, Leon AR, Tavazzi L, Sun JP, Nihoyannopoulos P, Merlino J, Abraham WT, Ghio S, Leclercq C, Bax JJ, Yu CM, Gorcsan J 3rd, St John Sutton M, De Sutter J, Murillo J. Results of the Predictors of Response to CRT (PROSPECT) trial. Circulation. 2008 May 20;117(20):2608-16. doi: 10.1161/CIRCULATIONAHA.107.743120. Epub 2008 May 5. PMID 18458170
- [Background] Koos R, Neizel M, Schummers G, Krombach GA, Stanzel S, Gunther RW, Kelm M, Kuhl HP. Feasibility and initial experience of assessment of mechanical dyssynchrony using cardiovascular magnetic resonance and semi-automatic border detection. J Cardiovasc Magn Reson. 2008 Nov 4;10(1):49. doi: 10.1186/1532-429X-10-49. PMID 18983646
- [Background] Tsao J, Kozerke S, Boesiger P, Pruessmann KP. Optimizing spatiotemporal sampling for k-t BLAST and k-t SENSE: application to high-resolution real-time cardiac steady-state free precession. Magn Reson Med. 2005 Jun;53(6):1372-82. doi: 10.1002/mrm.20483. PMID 15906282
- [Background] RUSHMER RF, CRYSTAL DK, WAGNER C, ELLIS RM. Intracardiac impedance plethysmography. Am J Physiol. 1953 Jul;174(1):171-4. doi: 10.1152/ajplegacy.1953.174.1.171. No abstract available. PMID 13065515
- [Background] Salo RW, Wallner TG, Pederson BD. Measurement of ventricular volume by intracardiac impedance: theoretical and empirical approaches. IEEE Trans Biomed Eng. 1986 Feb;33(2):189-95. doi: 10.1109/TBME.1986.325890. No abstract available. PMID 3957369
- [Background] Kaye G, Edgar D, Mudawi T, Lippert M, Czygan G. Can transventricular intracardiac impedance measurement discriminate haemodynamically unstable ventricular arrhythmias in human? Europace. 2007 Feb;9(2):122-6. doi: 10.1093/europace/eul150. PMID 17272334
- [Background] Osswald S, Cron T, Gradel C, Hilti P, Lippert M, Strobel J, Schaldach M, Buser P, Pfisterer M. Closed-loop stimulation using intracardiac impedance as a sensor principle: correlation of right ventricular dP/dtmax and intracardiac impedance during dobutamine stress test. Pacing Clin Electrophysiol. 2000 Oct;23(10 Pt 1):1502-8. doi: 10.1046/j.1460-9592.2000.01502.x. PMID 11060870
- [Background] Fornwalt BK, Gonzales PC, Delfino JG, Eisner R, Leon AR, Oshinski JN. Quantification of left ventricular internal flow from cardiac magnetic resonance images in patients with dyssynchronous heart failure. J Magn Reson Imaging. 2008 Aug;28(2):375-81. doi: 10.1002/jmri.21446. PMID 18666147
- [Background] Fornwalt BK, Arita T, Bhasin M, Voulgaris G, Merlino JD, Leon AR, Fyfe DA, Oshinski JN. Cross-correlation quantification of dyssynchrony: a new method for quantifying the synchrony of contraction and relaxation in the heart. J Am Soc Echocardiogr. 2007 Dec;20(12):1330-1337.e1. doi: 10.1016/j.echo.2007.04.030. Epub 2007 Jul 23. PMID 17643956